CLINICAL TRIAL: NCT01821963
Title: Telaprevir in Combination With Standard of Care in Hepatitis C Genotype 1 Infection in Patients With Hepatocellular Carcinoma Awaiting Liver Transplantation
Brief Title: Telaprevir Plus Standard of Care (SOC) in HCV Associated Hepatocellular Carcinoma (HCC)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Low referral rate due to new therapeutic options.
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012-0977
Record Dates: First submitted 2013-03-27; First posted 2013-04-01 (Estimated); Results first posted 2015-03-06 (Estimated); Last update posted 2020-09-24 (Actual); Status verified 2020-09

CONDITIONS: Infection
Keywords: Infection; Hepatitis C Genotype 1 Infection; Hepatitis C virus; HCV; Hepatocellular Carcinoma; HCC; Liver Transplantation; Pegylated Interferon Alfa 2a; PegIFN alfa-2a; Ribavirin; RBV; Telaprevir; Incivek; Antiviral drugs
MeSH Terms: conditions — Infections; Hepatitis C; Carcinoma, Hepatocellular | interventions — peginterferon alfa-2a; Ribavirin; telaprevir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pegylated Interferon Alfa 2a + Ribavirin + Telaprevir (Experimental): Triple combination with Telaprevir, PegIFN alfa-2a and Ribavirin administered for 12 weeks, followed by dual therapy with PegIFN alfa-2a and Ribavirin. Dual therapy continued for 48 weeks of total duration of therapy, as standard of care treatment for cirrhotic patients, or until day of transplantation, whichever comes first. Starting doses for standard of care pegylated interferon (PegIFN) alfa-2a 180 mcg subcutaneously once weekly, for ribavirin (RBV) 1,000 mg orally daily (< 75 kg) and 1,200 mg orally daily (≥ 75 kg), and for telaprevir 750 mg taken orally 3 times a day.
  Interventions: Drug: Pegylated Interferon Alfa 2a; Drug: Ribavirin; Drug: Telaprevir

INTERVENTIONS:
Drug: Pegylated Interferon Alfa 2a — Starting dose: 180 mcg subcutaneously once weekly.
  Other Names: PegIFN
Drug: Ribavirin — Starting dose: 1,000 mg by mouth daily.
Drug: Telaprevir — Starting dose: 750 mg by mouth 3 times a day.
  Other Names: Incivek

SUMMARY:
The goal of this clinical research study is to learn if the antiviral combination of telaprevir, pegylated Interferon Alfa 2a (PegIFN alfa-2a) and ribavirin (RBV) can prevent the virus from coming back after the liver transplant.

Telaprevir, PegIFN alfa-2a, and RBV are different antiviral drugs that work in combination at different stages of the HCV infection to stop the virus.

DETAILED DESCRIPTION:
Study Drug Administration:

If you are found to be eligible to take part in this study, you will take telaprevir 3 times a day. You will take RVB by mouth 2 times a day. You will receive PEGIFN alfa-2a by an injection under the skin 1 time a week.

Study Visits:

On the first day you take the study drug:

* You will have an eye exam performed by the study doctor.
* You will have a physical exam, including measurement of your vital signs (blood pressure, heart rate, temperature, and breathing rate).
* Blood (about 2 teaspoons) will be drawn for routine tests and to check for the hepatitis virus.
* You will be asked about any drugs you are taking or side effects you may be having.

Every Week while you are on study:

* You will have a physical exam, including measurement of your vital signs.
* Blood (about 2 teaspoons) will be drawn for routine tests and to check for the hepatitis C virus. If part of the blood sample is left over after the Hepatitis C testing, it will be stored in the laboratory as a back-up sample, in case the original samples get lost. This sample may also be used to check if the Hepatitis C virus has become resistant to the study drug. No extra blood will be drawn for this storage.
* You will be asked about any drugs you are taking or side effects you may be having.
* At Weeks 12, 24, 36, and 42, urine will be collected to check for infection and any other side effects to the drugs.

If you can become pregnant, you will have a urine pregnancy test every 4 weeks

Length of Treatment:

You may continue receiving the antiviral therapy for up to 48 weeks, as long as the doctor thinks it is in your best interest. You will no longer be able to take the study drug if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

Your participation on the study will be over after the follow-up visits.

Follow-Up Visits:

Beginning the day after you stop taking antiviral therapy (or the day of transplantation, whichever comes first), you will have up to 24 weeks of follow-up testing performed. About 4 and 20 weeks after your last dose:

* You will have a physical exam, including measurement of your vital signs.
* Blood (about 2 teaspoons) will be drawn for routine tests and to check for the hepatitis C virus.
* You will be asked about any side effects you may be having.
* At week 4 only, urine will be collected to check for infection and any other side effects to the drugs.

This is an investigational study. Telaprevir, PegIFN alfa-2a, and RBV are all FDA approved and commercially available for the treatment of HCV infection. The use of these drugs in preventing the HCV infection is investigational.

Up to 40 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females aged ≥ 18 and ≤ 70 years
2. Detectable Hepatitis C Virus ribonucleic acid (HCV-RNA) in serum
3. HCV genotype 1 infection
4. Child-Pugh-Turcotte (CPT) score < 7 and Model for End-Stage Liver Disease (MELD) score < 18
5. PegIFN alfa-2a/RBV-naïve or previously treated patients (partial responders, null responders and relapsers)
6. Hepatocellular carcinoma within transplant criteria in the United Network for Organ Sharing (UNOS) Region IV:

   1. Single lesion up to 6 cm, or
   2. Two or three lesions with largest no greater than 5 cm and the total tumor diameter no greater than 9 cm
7. Listed for liver transplantation
8. Willingness to give written consent and agree to double contraception

Exclusion Criteria:

1. Decompensated cirrhosis
2. Baseline platelet count less than 35,000/µL
3. Baseline hemoglobin level less than 10 g/dL
4. Baseline absolute neutrophil count less than 750/mm3
5. Baseline creatinine clearance < 50 mL per min.
6. Women with a positive pregnancy test at baseline or men whose female partners are pregnant or are contemplating pregnancy
7. Intolerance or contraindications to PegIFN alfa-2a/RBV use per standard treatment guidelines

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2013-04; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harrys A. Torres, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: April 2013 to February 2014. All recruitment done at The University of Texas MD Anderson Cancer Center.
Pre-assignment Details: Study terminated early due to changes in research, alternate therapeutic treatment options.
Period: Overall Study
Arm/Group | Pegylated Interferon Alfa 2a + Ribavirin + Telaprevir
Started | 1
Completed | 0
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: Study terminated with one participant, no analysis performed.
Arm/Group | Pegylated Interferon Alfa 2a + Ribavirin + Telaprevir
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Undetectable Viral Load 12 Weeks Post-transplant
Description: The primary endpoint is number of participants with undetectable viral load at 12 weeks post-transplant (Post-transplant virological response, (PTVR)) which is defined as undetectable Hepatitis C Virus ribonucleic acid (HCV-RNA) 12 weeks after liver transplantation). In order to have undetectable HCV RNA viral load after transplant, participants need to have undetectable viral load before the liver transplant.
  Response rate based on the modified intent-to-treat (ITT) population where ITT population is defined as those patients who have achieved an undetectable HCV-RNA level before the transplant. If patients drop out the study early due to severe toxicity or treatment failure including treatment-related death, they will be counted as non-responders when evaluating the response rate.
Time Frame: 12 weeks post-transplant, up to 48 weeks for overall monitoring
Population: Study terminated early with one participant. No analysis possible.
Arm/Group | Pegylated Interferon Alfa 2a + Ribavirin + Telaprevir
Number analyzed (Participants) | 0

2. Secondary Outcome: Sustained Virological Response (SVR)
Description: Sustained virological response (SVR) defined as a single undetectable HCV-RNA measurement 12 weeks after the 48-week treatment period for those still waiting for transplantation. The treatment duration will be summarized with descriptive statistics. Additional analyses based on evaluable patients also conducted regarding the PTVR response rate. The evaluable patients are defined as those patients who complete at least 16 weeks of treatment and have the 12 weeks post-transplant response measurement. The rate will also be computed stratified by the HCV treatment time (i.e., the 48-week HCV treatment versus less than 48 week HCV treatment) considering the different times under HCV. The SVR rate will be estimated, along with the exact 95% confident interval.
Time Frame: 60 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse event data collection through baseline HCV therapy through the Safety Follow-up Visit, with the last visit 24 weeks post end-of-treatment (or following liver transplantation). Overall active study period: May 1 to June 21, 2013.
Description: Study terminated early without a treatment completion.
Arm/Group | Pegylated Interferon Alfa 2a + Ribavirin + Telaprevir
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pegylated Interferon Alfa 2a + Ribavirin + Telaprevir (N=1)
Retinopathy (Eye disorders) | 1 (1)
Nonoliguric acute kidney injury (Renal and urinary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes